CLINICAL TRIAL: NCT06470763
Title: A First-in-human, Open-label, Multicenter Phase I/II Study to Evaluate the Safety and Anti-tumor Activity of ANV600 As Single Agent and in Combination with Pembrolizumab in Participants with Advanced Solid Tumors (EXPAND-1)
Brief Title: A Study Evaluating ANV600 Single Agent or in Combination with Pembrolizumab in Participants with Advanced Solid Tumors (EXPAND-1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anaveon AG (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANV600-001; EXPAND-1 (Other: ANAVEON AG); KEYNOTE-F78 (Other: Merck Sharp & Dohme LLC); MK-3475-F78 (Other: Merck Sharp & Dohme LLC); 2023-509633-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ANV600 single agent (Experimental)
  Interventions: Drug: ANV600
- ANV600 in combination with pembrolizumab (KEYTRUDA®) (Experimental)
  Interventions: Drug: ANV600 + pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: ANV600 — ANV600 administered by intravenous (IV) infusion
  Arms: ANV600 single agent
Drug: ANV600 + pembrolizumab (KEYTRUDA®) — ANV600 administered by intravenous (IV) infusion pembrolizumab (KEYTRUDA®) administered by intravenous (IV) infusion
  Arms: ANV600 in combination with pembrolizumab (KEYTRUDA®)

SUMMARY:
The purpose of study ANV600-001 is to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, immunogenicity and antitumor activity of ANV600 administered as a single agent or in combination with pembrolizumab in adult participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* The participant provides written informed consent for the trial;
* Life-expectancy ≥ 3 months;
* Able to comply with the Protocol as judged by the Investigator;
* ≥ 18 years of age on day of signing informed consent;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* Measurable disease per RECIST v1.1;
* Adequate organ function, defined as:

  * Absolute neutrophil count (ANC) ≥1200/µL;
  * Platelet count ≥100 000/µL;
  * Hemoglobin ≥9.0 g/dL;
  * Measured or calculated creatinine clearance ≥50 mL/min;
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases);
  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN;
* Phase I: Advanced unresectable or metastatic solid tumors for which no standard of care treatments are available, or participants who cannot tolerate such treatment;
* Phase II: Tumor-specific cohorts in adult participants with advanced solid tumors:

  * Cohort A: Unresectable Stage III or Stage IV cutaneous melanoma (excl. mucosal and uveal), which has progressed on/after treatment with a PD-1/L1 checkpoint inhibitor;
  * Cohort B: Unresectable or metastatic squamous or non-squamous non-small cell lung cancer (NSCLC) not eligible for an approved targeted therapy, which has progressed on/after treatment with a PD-1/L1 checkpoint inhibitor;
  * Cohort C: Recurrent and/or unresectable/metastatic head and neck squamous cell carcinoma (HNSCC) (except nasopharyngeal carcinoma), after platinum failure and a PD-1/L1 checkpoint inhibitor.

Additional inclusion criteria apply as per study protocol

Exclusion criteria

* Pancreatic cancer (e.g. PDAC) (Phase I only);
* Primary or secondary adrenal insufficiency (Phase I only);
* History of allergic reactions attributed to any of the excipients of ANV600, such as sucrose, histidine or polysorbate 80. For combination only: severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients;
* Investigational agent (including investigational device) within 4 weeks or an interval of five half-lives of the respective investigational agent prior to study Day 1, whichever is shorter;
* Received IL-2 or IL-2 analogues as anti-cancer therapy within 18 months prior to study Day 1 (except IL-2 given in combination with cell therapy [e.g. TILs]);
* Not recovered (i.e. ≤ Grade 1 at baseline) from AEs resulting from prior immunotherapies with the following exceptions:

  1. Autoimmune AEs controlled by replacement therapy (e.g., hypothyroidism, adrenal insufficiency)
  2. Vitiligo or alopecia
  3. Psoriasis;
* Received prior systemic anti-cancer therapy including investigational agents within 4 weeks (could consider shorter interval for kinase inhibitors or other short half-life drugs) prior to treatment; Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
* For combination only: Have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g.CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher irAE;
* Active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment;
* Additional malignancy that is progressing or has required active treatment within the past 3 years;
* Active autoimmune disease that has required systemic treatment in the past 2 years;
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug;
* Allogeneic tissue/solid organ or stem cell transplant;
* History of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease;
* Active infection requiring systemic therapy;

Additional exclusion criteria apply per study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Phase I dose escalation: Incidence of Dose Limiting Toxicities (DLT) with ANV600 single agent and in combination with pembrolizumab combination with pembrolizumab | Day 1 up to 24 months
Phase I dose escalation: Frequency and severity of treatment-emergent adverse events (TEAEs) with ANV600 and in combination with pembrolizumab | Day 1 up to 24 months
Phase II: Objective Response Rate (ORR) using RECIST v1.1 | Day 1 up to 24 months
Phase II: Duration of Response (DOR) using RECIST v1.1 | Day 1 up to 24 months

SECONDARY OUTCOMES:
Phase I Dose escalation: Serum concentration of ANV600 following a single dose and after repeated dosing | Day 1 up to 24 months
Phase I Dose escalation: Immunogenicity as indicated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (nAb) | Day 1 up to 24 months
Phase I Dose escalation: Objective response rate (ORR) using RECIST v1.1 | Day 1 up to 24 months
Phase I Dose escalation: Duration of response (DOR) using RECIST v1.1 | Day 1 up to 24 months
Phase II: Progression-free survival (PFS) | Day 1 up to 24 months
Phase II: Overall Survival (OS) | Day 1 up to 24 months
Phase II: Frequency and severity of treatment-emergent adverse events (TEAEs) with ANV600 and in combination with pembrolizumab | Day 1 up to 24 months
Phase II: PK parameters based on ANV600 serum levels following a single dose and after repeated dosing | Day 1 up to 24 months
Phase II: Immunogenicity as indicated by the incidence of antidrug antibodies (ADA) and neutralizing antibodies (nAb) | Day 1 up to 24 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (3):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (4):
  - Institut Bergonie, Bordeaux
  - CEPCM - AP-HM Hopital de la Timone, Marseille
  - Oncopole Claudius Regaud, Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Krankenhaus Nordwest - Institut für Klinisch-Onkologische Forschung (IKF), Frankfurt
  - Universitaetsmedizin der Johannes Gutenberg - Universitaet Mainz, Mainz
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, Netherlands
- Spain (4):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - START Madrid CIOCC, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - INCLIVA Foundation, Valencia
- Switzerland (2):
  - Ente Ospedaliero Cantonale - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Cantonal Hospital St Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Undecided